CLINICAL TRIAL: NCT07111637
Title: Artificial Intelligence-Assisted Magnetic Resonance Imaging for Quality, Efficiency and Equity in the National Health Service (NHS) Care of Multiple Sclerosis
Acronym: AssistMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: icometrixLeuven (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Worktribe 8529379; AI_AWARD02608 (Other Grant/Funding Number: National Institute for Health & Care Research (NIHR UK))
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiological reading by a neuroradiologist assisted by icobrain ms. (Experimental): icobrain ms Artificial Intelligence (AI) assistive software
  Interventions: Device: AI software
- Radiological reading by a neuroradiologist (No Intervention): Standard of Care

INTERVENTIONS:
Device: AI software — icobrain ms is an Artificial Intelligence (AI)-assistive software which quantifies brain Magnetic Resonance Imaging (MRIs) and summarises clinically relevant findings for patients with Multiple Sclerosis in structured electronic radiological reports and annotated images.
  Arms: Radiological reading by a neuroradiologist assisted by icobrain ms.

SUMMARY:
Multiple Sclerosis (MS) is a long-term disease that affects over 150,000 people in the UK. Starting treatment early is important for managing Multiple Sclerosis (MS). It is also essential to monitor the treatment to see if it is working and to switch treatments if needed.

Magnetic resonance imaging (MRI) is the only accepted tool to monitor how well the treatment is working. Current evaluation of brain Magnetic resonance imaging (MRI) scans requires visual inspection, of which sensitivity is degraded by human, and technical factors, such as lack of time, fatigue of radiologists, and lack of standardization of image acquisition protocols across the National Health Service (NHS). MRI-readings can be significantly enhanced by artificial intelligence (AI)-assistive software. Evidence suggests the rate of new lesion detection to be 3 - 4 times higher when using assistive software compared to visual inspection of MRI scans.

In this study, an Artificial Intelligence (AI) software called "icobrain ms." developed by the company "icometrix" (Leuven, Belgium) is tested. This tool helps track MS by measuring changes in the brain using MRI scans. The AI can highlight problem areas and create reports that doctors can use to make better decisions about participants' treatment. The aim of the study is to prove that icobrain ms can be used to assist the neuro-radiologist with their visual assessment of MRI scans by a radiologist, and that it will help clinicians make more informed decisions about participants' current MS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Isolated Syndrome suggestive of demyelination (CIS) or definitive diagnosis of MS.
* Undergoing MRI head investigation.
* On an MS DMT pathway.
* Access to a smartphone, tablet or computer.

Exclusion Criteria:

* patients with Multiples Sclerosis participating in a randomised controlled CTIMP (participating in a single arm study may be included, provided this is in line with the other protocol).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1336 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical usefulness of icobrain ms by evaluating the detection of disease activity (as defined by new/expanding lesions). | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.isrctn.com/ISRCTN99207647